CLINICAL TRIAL: NCT04854941
Title: Efficacy of Probiotics (Lactobacillus Rhamnosus, Bifidobacterium Bifidum, Bifidobacterium Longum Subsp. Infantis and Bifidobacterium Longum) in the Treatment of Hospitalised Patients With Novel Coronavirus Infection
Brief Title: Efficacy of Probiotics in the Treatment of Hospitalised Patients With Novel Coronavirus Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROCOV-19-2020
Record Dates: First submitted 2021-04-07; First posted 2021-04-22 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-04

CONDITIONS: Coronavirus Infection
Keywords: Novel Coronavirus Infection; Probiotics; Lactobacillus; Bifidobacterium; Clinical outcomes; C.difficile; Diarrhea; Liver; mortality
MeSH Terms: conditions — Coronavirus Infections; Diarrhea | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (PRO) (Experimental): 99 patients with COVID-19 infection who have been supplemented with a Lactobacillus and Bifidobacterium containing probiotic in addition to standard regimen (oxygen support, antiviral, antibacterial, anticoagulant, anticytokine (tocilizumab and olokizumab) drugs and dexamethasone treatment according to indications and contraindications)
  Interventions: Other: Probiotics
- Control group (CON) (No Intervention): 101 patients with COVID-19 infection who have been treated with standard regimen only (oxygen support, antiviral, antibacterial, anticoagulant, anticytokine (tocilizumab and olokizumab) drugs and dexamethasone treatment according to indications and contraindications)

INTERVENTIONS:
Other: Probiotics — Probiotics (10^9 CFU of each strain: Lactobacillus rhamnosus PDV 1705, Bifidobacterium bifidum PDV 0903, Bifidobacterium longum subsp. infantis PDV 1911 and Bifidobacterium longum PDV 2301) 3 times per day in addition to standard treatment regimen for 2 weeks
  Arms: Probiotics group (PRO)

SUMMARY:
The treatment of the new coronavirus infection (COVID-19) and COVID-19-associated diarrhoea and liver injury remains challenging. Optimizing treatment approaches for COVID-19 remains an issue. It is assumed, that changes in composition of intestinal microbiota is closely related to a change in the regulation of the immune response in the lungs in patients with COVID-19. These gut microbiota changes in combination with antibiotic prescription during the treatment increase the risk of antibiotic-associated diarrhea and C. difficile infection as well as worse clinical outcomes in these patients. Probiotics are useful for restoring the human gut microbiome and increasing anti-inflammatory response also. Despite the variety of uses of probiotics, there is still insufficient data on the clinical efficacy of including probiotics in the treatment of patients with COVID-19 infection.

DETAILED DESCRIPTION:
A randomized controlled open-label study approved by the local ethical committee. The study included patients with COVID-19 admitted to the T.M. Tareev Clinic of Internal Diseases of I.M. Sechenov First Moscow State Medical University in whom the disease was confirmed using polymerase chain reaction on nasopharyngeal and oropharyngeal swabs to detect severe acute respiratory syndrome-related coronavirus 2 (SARS-COV-2). The study was conducted from December 2020 to March 2021 and included participants in the age range from 18 to 75 years.

The exclusion criteria were age over 75 years or under 18 years, consumption of probiotics for 3 months prior to admission, history of intolerance to probiotics or their components, refusal to participate and sign informed consent, pregnancy or breastfeeding, cancer or mental illness, and severe renal (glomerular filtration rate less than 50 mL/min) or hepatic (equivalent to cirrhosis class B or C on the Child-Pugh scale) dysfunction at the time of admission.

Patients who prematurely discontinued the consumption of probiotics for reasons not related to the development of side effects were excluded from the study.

The patients were randomised to the probiotics group (PRO group) or the control group (CON group). Patients in the PRO group received probiotics containing ~109 colony forming units (CFU) of Lactobacillus rhamnosus PDV 1705, ~109 CFU of Bifidobacterium bifidum PDV 0903, ~109 CFU of B. longum subsp. infantis PDV 1911, and ~109 CFU of B. longum PDV 2301 three times a day during the hospital stay but for no more than 14 days (PDV is the commercial letter designation of the bacterial strains). The end point of the trial was day 14 of hospitalisation or the day of the patient's discharge or death, whichever occurred earlier.

The control group consisted of patients who did not receive probiotics. Patients in both the groups also received dexamethasone and antiviral (favipiravir and/or riamilovir), antibacterial, anticoagulant (enoxaparin in most cases; rivaroxaban and dabigatran were used much less frequently), and anticytokine (tocilizumab or/and olokizumab) drugs according to indications and contraindications.

Death from any cause was considered the primary outcome. Duration of hospitalisation, total duration of the disease, incidence of admission to intensive care unit, need for oxygen support or mechanical ventilation, and changes in the values of key biomarkers were considered the main secondary outcomes. The duration of diarrhoea [loose or watery stools or an increase in the frequency of bowel movements (more than three times per day)] and incidence of hospital-acquired diarrhoea as well as the progression of pre-existing liver injury and onset of liver injury were considered additional secondary outcomes. Liver injury was determined through the presence of abnormalities in any of the main liver test findings (serum alanine transaminase, aspartate transaminase, alkaline phosphatase, gamma-glutamyl transferase, total bilirubin, and albumin levels).

The volume of the affected lungs was measured using chest computed tomography (CT); it included the sum of ground glass and consolidation volumes.

Results are presented as the median [interquartile range]. The groups were compared using Mann-Whitney test for continuous data and chi-square test for categorical data. Wilcoxon test was used to assess the changes in continuous biomarker values. Mortality was assessed using the Kaplan-Meier estimator and Cox's test. A p value ≤0.05 was considered the criterion for significance. Statistical calculations were performed using "Statistica 10" soft (TIBCO Software inc, Palo Alto, CA)

ELIGIBILITY:
Inclusion Criteria:

* patients with COVID-19 infection confirmed by polymerase chain reaction of nasopharyngeal and oropharyngeal swabs to the causative agent of this infection
* age from 18 to 75 years old from December 2020 to April 2021

Exclusion Criteria:

* the patient's decision to withdraw from the study
* refusing to take the probiotic for a reason not related to the development of side effects.

Non-inclusion criteria:

* age over 75 years old or under 18 years old,
* taking probiotics for 3 months prior to admission
* history of intolerance to probiotics or their components
* refusal to participate and sign informed consent
* pregnancy or breastfeeding
* presence of cancer or psychoemotional disorders
* renal failure at the time of admission (glomerular filtration rate less than 50 ml / min)
* hepatic failure at the time of admission (equivalent to cirrhosis class B or C on the Child-Pugh scale)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Mortality | During hospitalization (Since the first day of hospitalization to the day of the patient's discharge)
  The number of died patients during hospitalization

SECONDARY OUTCOMES:
Duration of hospitalization | Since the first day of hospitalization to the day of the patient's discharge
  The number of days patients stayed at hospital
Total duration of the disease | Since the first day of hospitalization to the day of the patient's discharge
  The number of days patients had complaints
Incidence of admission to intensive care unit | at the 14th day of hospitalization or at the day of the patient's discharge
  The number of patients admitted to the intensive care unit during hospitalization
Need for non-invasive ventilation | at the 14th day of hospitalization or at the day of the patient's discharge
  The number of patients requiring a non-invasive ventilation during hospitalization
Days of non-invasive ventilation | at the 14th day of hospitalization or at the day of the patient's discharge
  The number of days that patients had non-invasive ventilation during hospitalization
Need for invasive ventilation | at the 14th day of hospitalization or at the day of the patient's discharge
  The number of patients requiring an invasive ventilation during hospitalization
Changes in the values of C-reactive protein level in serum | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The values of C-reactive protein level (mg/L) in serum of the patients during hospitalization
Changes in the counts of white blood cells in blood test | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The counts of white blood cells (10^9/L) in blood test of the patients during hospitalization
Changes in the counts of neutrophils in blood test | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The counts of neutrophils (10^9/L) in blood test of the patients during hospitalization
Changes in the counts of lymphocytes | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The counts of lymphocytes (10^9/L) in blood test of the patients during hospitalization
Changes in the counts of platelets | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The counts of platelets (10^9/L) in blood test of the patients during hospitalization
Changes in the values of erythrocyte sedimentation rate in in blood test | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The values of erythrocyte sedimentation rate (mm/hr) in blood test of the patients during hospitalization
Changes in the values of creatinine level in serum | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The values of creatinine (μmol/l) level in serum of the patients during hospitalization
Changes in the values of alanine aminotransferase (ALT) level in serum | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The values of alanine aminotransferase (ALT) level (u/L) in serum of the patients during hospitalization
Changes in the values of aspartate aminotransferase level in serum | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The values of aspartate aminotransferase (AST) level (u/L) in serum of the patients during hospitalization
Changes in the values of albumen level in serum | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The values of albumen level (g/L) in serum of the patients during hospitalization
Changes in the values of total bilirubin level in serum | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The values of total bilirubin level (μmol/l) in serum of the patients during hospitalization
Changes in the values of lactate dehydrogenase level in serum | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The values of lactate dehydrogenase (LDH) level (u/l) in serum of the patients during hospitalization
Changes in the values of ferritin level in serum | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The values of ferritin level (μg/l) in serum of the patients during hospitalization
Changes in the values of fibrinogen level in serum | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The values of fibrinogen level (g/l) in serum of the patients during hospitalization
Changes in the values of potassium level in serum | at the first and at the 14th day of hospitalization (or at the first day and at day of the patient's discharge)
  The values of potassium level (mmol/l) in serum of the patients during hospitalization
Incidence of diarrhoea | at 14th day of hospitalization (or at the day of the patient's discharge)
  The number of patients with diarrhea (loose or watery stools or frequent bowel movements more than three times a day) during hospitalization
The duration of diarrhoea | at 14th day of hospitalization (or at the day of the patient's discharge)
  The number of days that the patients had diarrhea (loose or watery stools or frequent bowel movements more than three times a day)
The maximum volume of the affected lungs | at 14th day of hospitalization (or at the day of the patient's discharge)
  The volume of the affected lungs counted by the sum of ground glass and consolidation volumes (%) using chest computed tomography (CT)

CONTACTS AND LOCATIONS:
Locations (1):
- I.M. Sechenov First Moscow State Medical University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
The provision of data is prohibited by Local Ethical Committee and is possible upon receipt of an official request addressed to the principal investigator

REFERENCES:
- [Background] Madabhavi I, Sarkar M, Kadakol N. COVID-19: a review. Monaldi Arch Chest Dis. 2020 May 14;90(2). doi: 10.4081/monaldi.2020.1298. PMID 32498503
- [Background] Logunov DY, Dolzhikova IV, Zubkova OV, Tukhvatullin AI, Shcheblyakov DV, Dzharullaeva AS, Grousova DM, Erokhova AS, Kovyrshina AV, Botikov AG, Izhaeva FM, Popova O, Ozharovskaya TA, Esmagambetov IB, Favorskaya IA, Zrelkin DI, Voronina DV, Shcherbinin DN, Semikhin AS, Simakova YV, Tokarskaya EA, Lubenets NL, Egorova DA, Shmarov MM, Nikitenko NA, Morozova LF, Smolyarchuk EA, Kryukov EV, Babira VF, Borisevich SV, Naroditsky BS, Gintsburg AL. Safety and immunogenicity of an rAd26 and rAd5 vector-based heterologous prime-boost COVID-19 vaccine in two formulations: two open, non-randomised phase 1/2 studies from Russia. Lancet. 2020 Sep 26;396(10255):887-897. doi: 10.1016/S0140-6736(20)31866-3. Epub 2020 Sep 4. PMID 32896291
- [Background] Tariq R, Saha S, Furqan F, Hassett L, Pardi D, Khanna S. Prevalence and Mortality of COVID-19 Patients With Gastrointestinal Symptoms: A Systematic Review and Meta-analysis. Mayo Clin Proc. 2020 Aug;95(8):1632-1648. doi: 10.1016/j.mayocp.2020.06.003. Epub 2020 Jun 10. PMID 32753138
- [Background] Kumar A, Arora A, Sharma P, Anikhindi SA, Bansal N, Singla V, Khare S, Srivastava A. Gastrointestinal and hepatic manifestations of Corona Virus Disease-19 and their relationship to severe clinical course: A systematic review and meta-analysis. Indian J Gastroenterol. 2020 Jun;39(3):268-284. doi: 10.1007/s12664-020-01058-3. Epub 2020 Aug 4. PMID 32749643
- [Background] Rokkas T. Gastrointestinal involvement in COVID-19: a systematic review and meta-analysis. Ann Gastroenterol. 2020 Jul-Aug;33(4):355-365. doi: 10.20524/aog.2020.0506. Epub 2020 Jun 6. PMID 32624655
- [Background] Zarifian A, Zamiri Bidary M, Arekhi S, Rafiee M, Gholamalizadeh H, Amiriani A, Ghaderi MS, Khadem-Rezaiyan M, Amini M, Ganji A. Gastrointestinal and hepatic abnormalities in patients with confirmed COVID-19: A systematic review and meta-analysis. J Med Virol. 2021 Jan;93(1):336-350. doi: 10.1002/jmv.26314. Epub 2020 Jul 27. PMID 32681674
- [Background] Suresh Kumar VC, Mukherjee S, Harne PS, Subedi A, Ganapathy MK, Patthipati VS, Sapkota B. Novelty in the gut: a systematic review and meta-analysis of the gastrointestinal manifestations of COVID-19. BMJ Open Gastroenterol. 2020 May;7(1):e000417. doi: 10.1136/bmjgast-2020-000417. PMID 32457035
- [Background] Sultan S, Altayar O, Siddique SM, Davitkov P, Feuerstein JD, Lim JK, Falck-Ytter Y, El-Serag HB; AGA Institute. Electronic address: ewilson@gastro.org. AGA Institute Rapid Review of the Gastrointestinal and Liver Manifestations of COVID-19, Meta-Analysis of International Data, and Recommendations for the Consultative Management of Patients with COVID-19. Gastroenterology. 2020 Jul;159(1):320-334.e27. doi: 10.1053/j.gastro.2020.05.001. Epub 2020 May 11. PMID 32407808
- [Background] Wang H, Qiu P, Liu J, Wang F, Zhao Q. The liver injury and gastrointestinal symptoms in patients with Coronavirus Disease 19: A systematic review and meta-analysis. Clin Res Hepatol Gastroenterol. 2020 Oct;44(5):653-661. doi: 10.1016/j.clinre.2020.04.012. Epub 2020 May 12. PMID 32418852
- [Background] Mao R, Qiu Y, He JS, Tan JY, Li XH, Liang J, Shen J, Zhu LR, Chen Y, Iacucci M, Ng SC, Ghosh S, Chen MH. Manifestations and prognosis of gastrointestinal and liver involvement in patients with COVID-19: a systematic review and meta-analysis. Lancet Gastroenterol Hepatol. 2020 Jul;5(7):667-678. doi: 10.1016/S2468-1253(20)30126-6. Epub 2020 May 12. PMID 32405603
- [Background] Bottari B, Castellone V, Neviani E. Probiotics and Covid-19. Int J Food Sci Nutr. 2021 May;72(3):293-299. doi: 10.1080/09637486.2020.1807475. Epub 2020 Aug 12. PMID 32787470
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Spigaglia P. COVID-19 and Clostridioides difficile infection (CDI): Possible implications for elderly patients. Anaerobe. 2020 Aug;64:102233. doi: 10.1016/j.anaerobe.2020.102233. Epub 2020 Jun 25. PMID 32593567
- [Background] d'Ettorre G, Ceccarelli G, Marazzato M, Campagna G, Pinacchio C, Alessandri F, Ruberto F, Rossi G, Celani L, Scagnolari C, Mastropietro C, Trinchieri V, Recchia GE, Mauro V, Antonelli G, Pugliese F, Mastroianni CM. Challenges in the Management of SARS-CoV2 Infection: The Role of Oral Bacteriotherapy as Complementary Therapeutic Strategy to Avoid the Progression of COVID-19. Front Med (Lausanne). 2020 Jul 7;7:389. doi: 10.3389/fmed.2020.00389. eCollection 2020. PMID 32733907
- [Result] Ivashkin V, Fomin V, Moiseev S, Brovko M, Maslennikov R, Ulyanin A, Sholomova V, Vasilyeva M, Trush E, Shifrin O, Poluektova E. Efficacy of a Probiotic Consisting of Lacticaseibacillus rhamnosus PDV 1705, Bifidobacterium bifidum PDV 0903, Bifidobacterium longum subsp. infantis PDV 1911, and Bifidobacterium longum subsp. longum PDV 2301 in the Treatment of Hospitalized Patients with COVID-19: a Randomized Controlled Trial. Probiotics Antimicrob Proteins. 2023 Jun;15(3):460-468. doi: 10.1007/s12602-021-09858-5. Epub 2021 Oct 13. PMID 34643888